CLINICAL TRIAL: NCT01801540
Title: The Effects of L-arabinose in a Meal on Glucose Metabolism in Healthy Men
Brief Title: The Effects of L-arabinose in a Meal in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, AAstrup, Dr.Med.Sci./Ph.D., University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-2-2010-095
Record Dates: First submitted 2013-02-27; First posted 2013-02-28 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Glucose Metabolism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 0% arabinose meal sucrose/starch (Experimental): A meal containing a bon with butter and marmalade, a cup cake, The and water
  Interventions: Dietary Supplement: L-arabinose - effect on glucose metabolism
- 5 % arabinose meal sucrose/starch (Other): A meal containing a bon with butter and marmalade, a cup cake, The and water
  Interventions: Dietary Supplement: L-arabinose - effect on glucose metabolism
- 10 % arabinose meal sucrose/starch (Other): A meal containing a bon with butter and marmalade, a cup cake, The and water
  Interventions: Dietary Supplement: L-arabinose - effect on glucose metabolism
- 0 % arabinose meal Starch (Other): A meal containing two bons with butter and cheese, The and water
  Interventions: Dietary Supplement: L-arabinose - effect on glucose metabolism
- 5 % arabinose meal starch (Other): A meal containing two bons with butter and cheese, The and water
  Interventions: Dietary Supplement: L-arabinose - effect on glucose metabolism
- 10 % arabinose meal starch (Other): A meal containing two bons with butter and cheese, The and water
  Interventions: Dietary Supplement: L-arabinose - effect on glucose metabolism

INTERVENTIONS:
Dietary Supplement: L-arabinose - effect on glucose metabolism — L-arabinose is mixed into the dough of the buns and cup cakes

SUMMARY:
The purpose of this study is to investigate the effect of a meal containing different doses of L-arabinose, on the intestinal sucrase activity after intake We measure this by measuring the glucose, insulin and c-peptide after meals. Other measurements are made (glucagon and GLP-1) to explain the correlations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* normal weight (BMI 18,5-25 kg/m2)
* 18-30 years of age

Exclusion Criteria:

* Not healthy,including those with diabetes Mellitus, high bloodpressure, dyslipidemia or a infectious diseases (hepatitis or HIV), gastrointestinal disorders
* Central adipositas (defined as waist circumference > 94 cm for european men)
* Daily intake of vitamins and minerals, 3 months before the trail starts and during the trail.
* elevated alcoholcunsumption(> 21 units af alcohol pr. week)
* take medicine
* Elite athlete with intensive training
* given bloddonation within the last 3 months
* smoking

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Glucose | -15, 0, 15, 30, 45, 60, 90, 120, 180 min
  Level of glucose over time, The AUC, the peak value and time to peak
Insulin | -15, 0, 15, 30, 45, 60, 90, 120, 180 min
  Level of insulin over time, the AUC, the peak value and time to peak
C-peptide | -15, 0, 15, 30, 45, 60, 90, 120, 180 min
  Level of c-peptide over time, The AUC, the peak value and time to peak

SECONDARY OUTCOMES:
Glucagon | -15, 0, 15, 30, 45, 60, 90, 120, 180 min
  Level of glucagon over time, The AUC, the peak value and time to peak
GLP-1 | -15, 0, 15, 30, 45, 60, 90, 120, 180 min
  Level of GLP-1 over time, The AUC, the peak value and time to peak

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rikardt Andersen, MD, lector, Study Director — Unit of Nutrition 5711, Rigshospitalet, Blegdamsvej 9, 2100 København Ø